CLINICAL TRIAL: NCT04555447
Title: Gastrointestinal Tolerability to Increasing Doses of Agavins and Impact on Gut Microbiota, Fecal Metabolites, and Metabolic Biomarkers in Healthy and Obese Subjects
Brief Title: Gastrointestinal Tolerability to Agavins and Impact on Host-gut Microbiota-metabolism Interactions Modulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro De Investigación Y De Estudios Avanzados Del Instituto Politécnico Nacional-Unidad Irapuato (Other)
Collaborators: Centro de Estudios Cardiometabólicos S.C. (CESCAM) (Unknown); Inulina y Miel de Agave S.A. de C.V. (IMAG) (Unknown)
Responsible Party: Principal Investigator, Mercedes G. López, Professor, Centro De Investigación Y De Estudios Avanzados Del Instituto Politécnico Nacional-Unidad Irapuato
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CINVESTAV-IRA-BYB-171018
Record Dates: First submitted 2020-08-28; First posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Obesity; Healthy
Keywords: Prebiotics; Agavins; Gastrointestinal tolerability; Obesity; Gut microbiota; SCFA; Fecal metabolites; Agave dietary fiber
MeSH Terms: conditions — Obesity | interventions — maltodextrin

STUDY DESIGN:
Intervention Model Description: Healthy and obese participants randomized into agavins (prebiotic fiber) or placebo group received the corresponding dietary supplement simultaneously
Who Masked: Participant, Investigator
Masking Description: A research assistant not involved in the study was responsible for the generation of each participant's code, and for providing codified bags with ready-to-use sachets of each dietary supplement with the corresponding dose. The clinical trial coordinator enrolled participants, and investigators and participants were blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy-agavins (Experimental): Agavins are branched neo-fructans and were supplemented for a 5-week dose-escalation period in lean participants
  Interventions: Dietary Supplement: Agavins (prebiotic fiber)
- Healthy-placebo (Placebo Comparator): Maltodextrin was used as placebo and supplemented for a 5-week dose-escalation period in lean participants
  Interventions: Dietary Supplement: Placebo
- Obese-agavins (Experimental): Agavins are branched neo-fructans that were supplemented for a 5-week dose-escalation period in obese participants
  Interventions: Dietary Supplement: Agavins (prebiotic fiber)
- Obese-placebo (Placebo Comparator): Maltodextrin was used as placebo and supplemented for a 5-week dose-escalation period in obese participants
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Agavins (prebiotic fiber) — Agavins contained in ready-to-use sachets were dissolved in water, and participants consumed the corresponding dose daily (2.5, 5.0, 7.0, 10 or 12 g) for 1 week, preferentially in the evening. Participants followed a 5-week dose-escalation intervention.
  Other Names: Agave inulin (Preventy)
  Arms: Healthy-agavins; Obese-agavins
Dietary Supplement: Placebo — Maltodextrin contained in ready-to-use sachets was dissolved in water, and participants consumed the corresponding dose daily (2.5, 5.0, 7.0, 10 or 12 g) for 1 week, preferentially in the evening. Participants followed a 5-week dose-escalation intervention.
  Other Names: Maltodextrin (Globe 10 IP)
  Arms: Healthy-placebo; Obese-placebo

SUMMARY:
Agavins are branched neo-fructans and prebiotic fiber found in Agave plants. In preclinical studies, agavins have demonstrated an effect in reversing metabolic disorders associated to overweight and obesity through the modulation of gut microbiota activity and composition, showing their interesting potential in the context of high obesity and cardiovascular diseases prevalence in Mexican population. However, current information about gastrointestinal adaptation and effects of agavins intake in humans is scarce. We hypothesized that increasing amounts of agavins up to 12 g/day, will be well tolerated by healthy and obese adult participants, but with differences between these groups, modulating gut microbiota activity and structure differentially, as well as the metabolic status after a 5-week dose-escalation intervention.

DETAILED DESCRIPTION:
Diet has dramatically changed over the past decades with increased consumption of high-fat, high-sugar, high-sodium processed and refined foods, but with low or very low fiber-rich products. Microbiota-accessible carbohydrates (MACs) found for example in dietary fiber have been recognized as crucial for the microbial ecosystem in the gut; the lack of these available carbohydrates depletes the microbial community, causing alterations in its composition and performance. Perturbations in the gut microbiota have been related with several diseases, so as reduction in dietary fiber has been linked with an increased risk for developing chronic diseases, namely cardiovascular and metabolic ones, such as obesity and type 2 diabetes. Mexico is the second country with the highest obesity rates worldwide, which represents a major national public health challenge. Interestingly, national nutrition surveys have found that Mexican adults consume less than half the dietary intake recommendation for fiber, along with an alarming statistic of 7 in 10 adults being overweight or obese.

A change in dietary patterns intended to achieve adequate nutrient intake, dietary fiber included, is one strategy that could help modify this nutrition trend in the country, but another accessible alternative is the supplementation of prebiotic fiber, thus increasing fiber consumption and avoiding gut microbiota alterations simultaneously. Prebiotics, such as fructans, are substrates selectively used by gut microbes, modifying their activity and/or community composition, and conferring health benefits to the host. Clinical research has demonstrated their impact in reducing body weight, fat mass, hyperlipidemia, etc. Agave prebiotics, also known as agavins, are fructan-type carbohydrates that possess a unique molecular structure and are extracted as a complex multi-disperse mixture presenting different degrees of polymerization and/or branching. Previously, agavins have shown to induce weight loss, a significant reduction in glucose and total cholesterol levels, and promotion of satiety-related hormones in overweight mice through the increment in short-chain fatty acids (SCFA) and specific modulation of gut microbiota; more recently, fecal metabolomics have revealed interesting microbial-derived metabolites, detected after agavins supplementation in mouse models that could induce a beneficial effect on host health, but more research is needed.

Experts have stated that differences in dietary fiber structure guide its degradation: which microbes can metabolize these substrates, and the effects in the microbial community that overall, impact health. Additionally, structural differences in prebiotic fibers like agavins, may cause specific gastrointestinal (GI) adaptation and tolerance which is of great importance to promote their consumption and in determining an ideal amount or dose to further explore their impact.

In this study we propose a double-blind, placebo controlled, parallel groups, dose-escalation trial, where lean and obese subjects were assigned to either agavins or placebo group for a 5-week dose-escalation period. We aim to evaluate the evolution of GI tolerability and compared the records between lean and obese participants (Mexican adults), the impact in gut microbiota composition and activity through the determination of short-chain fatty acids and fecal metabolites, and metabolic status, all of this after a short period of time proposed to induce adaptation to agavins intake.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age 30 - 60 years
* BMI ≥ 30 kg/m2
* Stable body weight for at least 1 month prior to the study

Exclusion Criteria:

* Type 1 and type 2 diabetes
* Hypothyroidism
* Currently following a weight loss diet or physical activity regime for the same purpose
* Weight loss >3 kg within 3 months before enrollment
* Use of prebiotics, probiotics, or dietary fiber supplements
* Long-term (and within the preceding month) use of antioxidants, omega-3, and omega-6 fatty acids supplements
* Strenuous exercise (>3 hours/week)
* Concomitant use of any medication influencing appetite, weight, metabolism
* Use of metformin
* Antibiotic use 1 week prior to the study
* Alcohol or substance abuse
* Diagnosis of neurological or psychiatric disorders, like anxiety, depression, Attention-Deficit/Hyperactivity Disorder (ADHD), schizophrenia
* Active smoker
* Alanine Transaminase (ALT) and Aspartate Aminotransferase (AST) enzymes concentration >2.5 times the highest limit value
* Creatinine >1.2 mg/dL
* Women: pregnancy or lactation
* Previous intestinal or bariatric surgery
* Heart, brain, or thyroid surgeries within the preceding 6 months
* History of liver or pancreatic disease
* History of renal failure
* Intestinal absorption disorder
* Inflammatory bowel disease
* Established cardiovascular disease
* Active or history of neoplasia within the preceding 5 years
* Chronic use of bulk laxatives and antacids

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2019-09-07 (Actual); Study Completion 2019-09-07 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal tolerability | 0-5 weeks
  Five gastrointestinal symptoms related to tolerability (flatulence, bloating, borborygmi, diarrhea, and abdominal pain) were assessed by a 10-cm Visual Analog Scale (VAS), guided by "no effect" (0 cm) , "moderate effect" (5 cm), and "worst effect possible" (10 cm). Participants rated their feelings 12 hours after taking their daily dose of dietary supplement, at the same time every day. All VAS were provided as printed material, one scale for each gastrointestinal symptom.

SECONDARY OUTCOMES:
Appetite and satiety subjective assessment | 0-5 weeks
  Appetite and satiety feelings were assessed by a 10-cm Visual Analog Scale (VAS). Appetite ratings were guided by "How hungry do you feel?" anchored by "I am not hungry at all" and "I have never been hungrier; I have to eat immediately". Satiety ratings were guided by "How satisfied do you feel?" anchored by "I feel my stomach completely empty" and "I cannot eat another bite". Participants rated their feelings 12 hours after taking their daily dose of dietary supplement, at the same time every day. Each VAS was provided as printed material.
Gut microbiota composition | 5 weeks
  Gut microbiota composition was assessed by 16S rRNA sequencing
SCFA production | 5 weeks
  Short-chain fatty acids (SCFA) production was determined in feces by Gas Chromatography-Flame Ionization Detector (GC-FID), and expressed as SCFA concentration (µmol/g)
Fecal metabolomics | 5 weeks
  Fecal metabolomics will be performed by Gas Chromatography-Mass Spectrometry (GC-MS) . Ordination methods and statistical dimension reduction techniques such as Principal Component Analysis (PCA), Partial Least Square-Discriminant Analysis (PLS-DA), as well as hierarchical clustering analysis will be implemented to explore and identify clusters of samples, groups.

OTHER OUTCOMES:
Assessment of metabolic markers | 0-5 weeks
  Exploratory assessment of the concentration of clinically relevant metabolic markers, such as glucose, triglycerides, total cholesterol, HDL-C, LDL-C, etc., expressed in mg/dL was performed.
Body weight determination | 0-5 weeks
  Body weight (kg) was assessed by an 8-electrode bioelectrical impedance medical analyzer.
Fat mass, fat-free mass, body water, and skeletal muscle mass determination | 0-5 weeks
  Fat mass, fat-free mass, body water, and skeletal muscle mass percentages was assessed by an 8-electrode bioelectrical impedance medical analyzer.

CONTACTS AND LOCATIONS:
Overall Officials: Mercedes G. López, PhD, Study Director — Centro de Investigación y de Estudios Avanzados del Instituto Politécnico Nacional-UI
Locations (2):
- Mexico (2):
  - Centro de Investigación y de Estudios Avanzados del Instituto Politécnico Nacional-Unidad Irapuato (CINVESTAV-UI), Irapuato, Guanajuato
  - Centro de Estudios Cardiometabólicos S.C. (CESCAM), Mexico City

IPD SHARING:
Plan to Share IPD: No
Results will be published in a peer-reviewed journal in the fields of dietetics and nutrition, with impact factor according to the Journal Citation Reports.

REFERENCES:
- [Background] Huazano-Garcia A, Shin H, Lopez MG. Modulation of Gut Microbiota of Overweight Mice by Agavins and Their Association with Body Weight Loss. Nutrients. 2017 Aug 23;9(9):821. doi: 10.3390/nu9090821. PMID 28832493
- [Background] Franco-Robles E, Lopez MG. Agavins Increase Neurotrophic Factors and Decrease Oxidative Stress in the Brains of High-Fat Diet-Induced Obese Mice. Molecules. 2016 Aug 2;21(8):998. doi: 10.3390/molecules21080998. PMID 27490526
- [Background] Huazano-Garcia A, Lopez MG. Agavins reverse the metabolic disorders in overweight mice through the increment of short chain fatty acids and hormones. Food Funct. 2015 Dec;6(12):3720-7. doi: 10.1039/c5fo00830a. Epub 2015 Sep 3. PMID 26333285
- [Background] Santiago-Garcia PA, Lopez MG. Agavins from Agave angustifolia and Agave potatorum affect food intake, body weight gain and satiety-related hormones (GLP-1 and ghrelin) in mice. Food Funct. 2014 Dec;5(12):3311-9. doi: 10.1039/c4fo00561a. PMID 25367106
- [Background] Garcia-Vieyra MI, Del Real A, Lopez MG. Agave fructans: their effect on mineral absorption and bone mineral content. J Med Food. 2014 Nov;17(11):1247-55. doi: 10.1089/jmf.2013.0137. Epub 2014 Jul 28. PMID 25069021
- [Background] Urias-Silvas JE, Cani PD, Delmee E, Neyrinck A, Lopez MG, Delzenne NM. Physiological effects of dietary fructans extracted from Agave tequilana Gto. and Dasylirion spp. Br J Nutr. 2008 Feb;99(2):254-61. doi: 10.1017/S0007114507795338. Epub 2007 Aug 22. PMID 17711612